CLINICAL TRIAL: NCT03119038
Title: Efficacy of Intraoperative Injections on Postoperative Pain Control During Total Hip Arthroplasty: A Prospective, Blinded, Randomized Controlled Study
Brief Title: Efficacy of Intraoperative Injections on Postoperative Pain Control During Total Hip Replacement
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator no longer actively pursuing this study.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brett Levine, MD, Associate Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORA-15101602
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis; Degenerative Joint Disease
Keywords: total hip; degenerative joint disease; osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Joint Diseases | interventions — Epinephrine; Bupivacaine; Ropivacaine; Ketorolac; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Medication Injection (Active Comparator): Intraoperative periarticular injection of 300 mg of 0.5% ropivacaine, 30 mg ketorolac, 200 mcg epinephrine, and 100 mcg clonidine in a 100 mL 0.9% saline solution
  Interventions: Drug: Ropivacaine; Drug: Ketorolac; Drug: Clonidine Injection
- Single Medication Injection (Active Comparator): Intraoperative periarticular injection of 30 mL of a 0.25% solution bupivacaine with epinephrine and 30 mL 0.25% bupivacaine without epinephrine
  Interventions: Drug: Bupivicaine + epinephrine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivicaine + epinephrine — Intraoperative periarticular injection of 30 mL of a 0.25% solution bupivacaine with epinephrine
  Arms: Single Medication Injection
Drug: Bupivacaine — Intraoperative periarticular injection of 30 mL of a 0.25% solution bupivacaine without epinephrine
  Arms: Single Medication Injection
Drug: Ropivacaine — Intraoperative periarticular injection of 300 mg of 0.5% ropivacaine
  Arms: Combination Medication Injection
Drug: Ketorolac — Intraoperative periarticular injection of 30 mg
  Arms: Combination Medication Injection
Drug: Clonidine Injection — Intraoperative periarticular injection of 100 mcg clonidine in a 100 mL 0.9% saline solution
  Arms: Combination Medication Injection

SUMMARY:
The purpose of this study is to clarify the efficacy of a multidrug versus single drug periarticular injection when only standard operative and postoperative pain management protocols used and the control group is exposed to what our investigators believe is the standard of care, single medication periarticular injection

DETAILED DESCRIPTION:
Study Objectives The intraoperative periarticular injection of 300 mg of 0.5% ropivacaine, 30 mg ketorolac, 200 mcg epinephrine, and 100 mcg clonidine in a 100 mL 0.9% saline solution will be compared to an injection of 30 mL of a 0.25% solution bupivacaine with ORA: 15101602-IRB01 Date IRB Approved: 3/16/2016 epinephrine and 30 mL 0.25% bupivacaine without epinephrine as an intraoperative periarticular joint injection protocol. The study's data collection timeline begins at the pre-operative clinic visit. Data collection continues through the patient's discharge after the surgical procedure and until the first year postoperative visit examination of joint range of motion and patient satisfaction questionnaires.

Primary Objectives:

The primary objective is to evaluate the efficacy of a multidrug versus bupivacaine intraoperative injection in decreasing total hip arthroplasty postoperative pain. To determine this, postoperative analgesic consumption will be collected for each patient and the value when converted to morphine equivalents will be compared between cohorts.

Analysis of morphine equivalent values at various postoperative time intervals (0-6 hours, 6-12 hours, 12-18, 18-24, then each postoperative day) and total morphine equivalent consumption for the entire length of stay will be performed between treatment cohorts.

Secondary Objectives:

To establish the improvement in postoperative pain relief provided by intraoperative periarticular injection of our multidrug protocol versus bupivacaine, other data points will be collected. The physical therapy milestones including time to first get out of bed, time to ambulation with or without assistance, time to climb stairs, and time to active straight leg raise will all be collected. The zero time point will be the end of the operation. Pain scale scores during physical therapy sessions with physiotherapists will also be recorded.

Resting visual analog scores for pain assessment will be collected as the patient representing their pain on a scale from 0 to 100 mm. The VAS values will be collected at various postoperative time values until discharge. The length of hospital stay will be collected as well. Opioid side effects will also be collected including over sedation, respiratory depression, urinary retention, and constipation. Other data collected will include operation time, wound complications, intraoperative blood loss, and postoperative drain output. At the 6 weeks postoperative visit, patient satisfaction questionnaires will be collected compared to preoperative visit values.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be male or female of any race
2. Ages 18-80 years old
3. Patients must have a primary hip arthroplasty by principal investigator or co-investigator

Exclusion Criteria

1. Allergy or intolerance to the study materials
2. Surgical intervention during the past month for the treatment of the painful joint or its underlying etiology
3. History of previous surgeries on the affected joint other ORA: 15101602-IRB01 Date IRB Approved: 3/16/2016 than arthroscopy (open surgeries)
4. History of or current substance abuse or addiction
5. History of or current psychiatric diagnosis
6. Failure in collecting a required data point during study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04-30 (Estimated); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Record narcotic usage, in morphine equivalents, during postoperative inpatient hospital stay. | From date of randomization until the date of hospital discharge or the date of 10 days after surgery, whichever date comes first
  Narcotic usage

SECONDARY OUTCOMES:
Record time to achieve physical therapy milestones during inpatient physical therapy | From date of randomization until the date of hospital discharge or the date of 10 days after surgery, whichever date comes first
  Time to achieve physical therapy milestones
Record VAS values during postoperative period | From date of randomization until the date of hospital discharge or the date of 10 days after surgery, whichever date comes first
  VAS values
Length of hospital stay | From date of randomization until the date of hospital discharge or the date of 10 days after surgery, whichever date comes first
  Length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No